CLINICAL TRIAL: NCT05913960
Title: the Mechanism of Accelerated Intermittent Theta Burst Stimulation for Rapid Treatment of Major Depressive Disorder Based on the Prefrontal Excitation-inhibition Balance Regulated by CAMKII Pathway
Brief Title: Accelerated Intermittent Theta-Burst Stimulation Ameliorate Major Depressive Disorder by Regulating CAMKII Pathway
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IITA20230315
Record Dates: First submitted 2023-03-16; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder; Major Depressive Disorder, Recurrent
Keywords: major depressive disoerder; first episode without medication; recurrent unmedicated
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo stimulation (Sham Comparator): The sham group of MDD will receive sham rTMS stimulation.
  Interventions: Device: sham stimulation
- accelerated intermittent theta burst stimulation (Active Comparator): Stimulation site: According to the localization of neural orientation navigation system, magnetic resonance data was read in Brainsight software, and three-dimensional brain reconstruction was carried out. The stimulation target was located in the coordinates of Montreal Neurological Institute (MNI), which was located in the left dorsolateral prefrontal cortex BA46(-44, 40, 29).The treatment intensity was 100% exercise threshold, and a TBS stimulus series was stimulated for 2 seconds, including 10 times of 3 intra plexus stimuli of 50Hz and 5Hz intraplexus stimuli, 10s of interval, repeated 60 times, that is, a total of 1800 pulses per treatment, 10 times a day, 50 minutes interval, a total of 18000 pulses per day, continuous for 5 days.
  Interventions: Device: accelerated intermittent theta burst stimulation
- high frequency stimulation (Active Comparator): Stimulation site: According to the localization of neural orientation navigation system, magnetic resonance data was read in Brainsight software, and three-dimensional brain reconstruction was carried out. The stimulation target was located in the coordinates of Montreal Neurological Institute (MNI), which was located in the left dorsolateral prefrontal cortex BA46(-44, 40, 29).Treatment intensity was 100% exercise threshold, continuous 10Hz stimulation, repeated 75 times, that is, 3000 pulses per treatment, 6 times a day, 50 minutes interval, a total of 18000 pulses per day, continuous stimulation for 5 days.
  Interventions: Device: high frequency stimulation

INTERVENTIONS:
Device: sham stimulation — The parameters in the sham arm will be as above with the internal randomization of the device internally switching to sham in a blinded fashion.
  Arms: Placebo stimulation
Device: accelerated intermittent theta burst stimulation — Participants in the active stimulation group will receive the accelerated intermittent TBS to left DLPFC. The L-DLPFC will be targeted utilizing the neuronavigation system. Stimulation intensity will be standardized at 90% of RMT.
  Stimulation will be delivered to the L-DLPFC using an NTK-TMS-II100 TMS device,is compatible with the Brainsight TMS navigation system.
  Arms: accelerated intermittent theta burst stimulation
Device: high frequency stimulation — Participants in the active stimulation group will receive the high frequnency stimulation to left DLPFC. The L-DLPFC will be targeted utilizing the neuronavigation system. Stimulation intensity will be standardized at 90% of RMT.
  Stimulation will be delivered to the L-DLPFC using an NTK-TMS-II100 TMS device,is compatible with the Brainsight TMS navigation system.
  Arms: high frequency stimulation

SUMMARY:
Major depressive disorder(MDD) is a complex and heterogeneous mental disorder. Repeated transcranial magnetic stimulation (rTMS), as a non-invasive neuroregulatory technique, has shown a promising function in the treatment of depression. Theta-burst transcranial magnetic stimulation (TBS) model significantly shortened the duration of physical therapy treatment, and iTBS under the accelerated model (The latter is referred to as aiTBS)showed promising therapeutic effect. However, whether aiTBS has a better and faster curative effect in the first untreated or recurrent unmedicated MDD patients and the mechanism of its alleviation of depressive symptoms remains unclarified. This project intends to verify changes in CAMKII levels, CAMKII molecules and GABA receptors in brain-derived exosomes in normal controls and patients who received sham, aiTBS and high-frequency (10Hz) stimulation respectively. Neuroimaging and TMS-EEG were used to pinpoint the target of stimulation and to record the changes of brain waves before and after treatment in real time. To clarify the neurobiological mechanism of aiTBS rapidly improving depression, and to provide a new strong evidence for clinical transcranial magnetic stimulation for accurate treatment of MDD patients.

ELIGIBILITY:
Inclusion Criteria:

* Sign a written informed consent to participate in the trial and receive treatment;
* Major depressive disorder diagnosis;
* Hamilton depression scale (HAMD - 24) 24 total score 20 points or more;
* First episode or recurrence of depression patients, not taking psychiatric drugs;
* The han nationality, right-handed;
* Junior high school or above;

Exclusion Criteria:

* Other organic mental disorders and mental retardation and other severe mental disorders;
* Infection, trauma, and autoimmune diseases or other possible interference test evaluation of disease;
* Alcohol and drug dependence or is being treated for a hormone drugs patients;
* Craniocerebral injury;
* Seizure or a family history of epilepsy;
* Pregnancy and lactation women;
* All landowners had a metal and MRI contraindications or MRI examination revealed abnormal brain structure.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Hamilton depression scale-24 | baseline
  Assessement of depressive status,a score of more than 35 May indicate severe depression; More than 20 points, may be mild or moderate depression; A score of less than 8 indicates no symptoms of depression
Hamilton depression scale-24 | 5days
  Assessement of depressive status,a score of more than 35 May indicate severe depression; More than 20 points, may be mild or moderate depression; A score of less than 8 indicates no symptoms of depression
Hamilton depression scale-24 | 4 weeks
  Assessement of depressive status,a score of more than 35 May indicate severe depression; More than 20 points, may be mild or moderate depression; A score of less than 8 indicates no symptoms of depression

SECONDARY OUTCOMES:
Change in the score of THINC-it. | Baseline
  THINC-it is a computerized cognitive screening tool that is designed to assess cognitive function in adults. THINC-it stands for "THINking Clearly," and it includes a series of brief tests that evaluate several cognitive domains, including attention, working memory, executive function, and processing speed. The tool is administered on a tablet or computer, and it takes approximately 20 minutes to complete.
Change in the score of THINC-it. | 5 days
  THINC-it is a computerized cognitive screening tool that is designed to assess cognitive function in adults. THINC-it stands for "THINking Clearly," and it includes a series of brief tests that evaluate several cognitive domains, including attention, working memory, executive function, and processing speed. The tool is administered on a tablet or computer, and it takes approximately 20 minutes to complete.
Change in the score of THINC-it. | 4 weeks
  THINC-it is a computerized cognitive screening tool that is designed to assess cognitive function in adults. THINC-it stands for "THINking Clearly," and it includes a series of brief tests that evaluate several cognitive domains, including attention, working memory, executive function, and processing speed. The tool is administered on a tablet or computer, and it takes approximately 20 minutes to complete.
Change in neuroimaging using functional magnetic resonance | Baseline
  Scanning functional magnetic resonance. Functional magnetic resonance imaging (fMRI) is a neuroimaging technique that is used to measure changes in brain activity by detecting changes in blood flow. In the context of major depression, fMRI has been used to study changes in brain function that may be associated with the condition. Research using fMRI in major depression has shown that there are alterations in the activity of certain brain regions in people with the condition. Specifically, fMRI studies have identified changes in the activity of the prefrontal cortex, the amygdala, and the hippocampus in people with major depression. Overall, fMRI has provided valuable insights into the neural mechanisms underlying major depression, and may help to inform the development of new treatments for the condition.
Change in neuroimaging using functional magnetic resonance | 5 days
  Scanning functional magnetic resonance. Functional magnetic resonance imaging (fMRI) is a neuroimaging technique that is used to measure changes in brain activity by detecting changes in blood flow. In the context of major depression, fMRI has been used to study changes in brain function that may be associated with the condition. Research using fMRI in major depression has shown that there are alterations in the activity of certain brain regions in people with the condition. Specifically, fMRI studies have identified changes in the activity of the prefrontal cortex, the amygdala, and the hippocampus in people with major depression. Overall, fMRI has provided valuable insights into the neural mechanisms underlying major depression, and may help to inform the development of new treatments for the condition.
Change of blood factor levels | baseline
  Factors carried by peripheral blood and exosomes(Calcium/calmodulin dependent kinase II, cyclic-AMP dependent protein kinase A,protein kinase C and so on ).
Change of blood factor levels | 5 days
  Factors carried by peripheral blood and exosomes(Calcium/calmodulin dependent kinase II, cyclic-AMP dependent protein kinase A,protein kinase C and so on ).
Change of blood factor levels | 4 weeks
  Factors carried by peripheral blood and exosomes(Calcium/calmodulin dependent kinase II, cyclic-AMP dependent protein kinase A,protein kinase C and so on ).
Change in electroencephalogram | baseline
  Electroencephalogram is collected from 64 electrodes. EEG can be used to identify patterns of brain activity that are associated with the condition and to inform treatment decisions. EEG can be a useful tool for identifying patterns of brain activity that are associated with MDD and for guiding treatment decisions. Neurofeedback and TMS are two approaches that have shown promise in the treatment of MDD. several parameters are analyzed to identify patterns of brain activity that may be associated with the condition. These parameters include: Alpha power, Beta power, Theta power, Delta power, Coherence, and more.
Change in electroencephalogram | 5 days
  Electroencephalogram is collected from 64 electrodes. EEG can be used to identify patterns of brain activity that are associated with the condition and to inform treatment decisions. EEG can be a useful tool for identifying patterns of brain activity that are associated with MDD and for guiding treatment decisions. Neurofeedback and TMS are two approaches that have shown promise in the treatment of MDD. several parameters are analyzed to identify patterns of brain activity that may be associated with the condition. These parameters include: Alpha power, Beta power, Theta power, Delta power, Coherence, and more.
Hamilton anxiety scale | baseline
  Assessement of anxious status.A total score of more than 29 May indicate severe anxiety; Over 21 points, there may be significant anxiety; More than 14 points, may have moderate anxiety; More than 7 points, may have mild anxiety; If the score is less than 7, there are no symptoms of anxiety
Hamilton anxiety scale | 5 days
  Assessement of anxious status.A total score of more than 29 May indicate severe anxiety; Over 21 points, there may be significant anxiety; More than 14 points, may have moderate anxiety; More than 7 points, may have mild anxiety; If the score is less than 7, there are no symptoms of anxiety
Hamilton anxiety scale | 4 weeks
  Assessement of anxious status.A total score of more than 29 May indicate severe anxiety; Over 21 points, there may be significant anxiety; More than 14 points, may have moderate anxiety; More than 7 points, may have mild anxiety; If the score is less than 7, there are no symptoms of anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang, China